CLINICAL TRIAL: NCT02475395
Title: A Clinical Study Evaluating Consumer Use of a New Device (TRAK) to Measure Sperm Concentration From Human Semen Samples, and Comparing TRAK Test Results With Laboratory Reference Method Testing
Brief Title: Study of the Consumer Use of a New Home Test to Measure Sperm Concentration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sandstone Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SD001
Record Dates: First submitted 2015-06-09; First posted 2015-06-18 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-09

CONDITIONS: Fertility, Male; Sub-Fertility, Male
Keywords: Male Fertility; Male Infertility; Fertility; Sperm; Sperm Concentration
MeSH Terms: conditions — Infertility, Male

ARMS (2):
- Donor/Tester Subjects (Experimental): Male subjects use the TRAK device to attain a measurement of sperm concentration from their semen specimen
  Interventions: Device: TRAK device
- Tester Only Subjects (Experimental): Male or female subjects use the TRAK device to attain a measurement of sperm concentration from another donor's semen specimen.
  Interventions: Device: TRAK device

INTERVENTIONS:
Device: TRAK device — Use of TRAK to attain sperm concentration measurement
  Other Names: Sperm Concentration

SUMMARY:
The objective of the study is to evaluate the agreement in measurement of sperm concentration in human semen between lay users with TRAK and a recognized reference method. The study will also include the measurement of matched samples by TRAK when tested by healthcare professionals trained in use of the TRAK device.

ELIGIBILITY:
Inclusion Criteria:

Subjects (Donor/Tester)

* Generally healthy (apart from fertility or reproductive care), ambulatory, and have absence of chronic conditions or treatments, except those related to fertility and reproductive care
* 20 - 50 years of age inclusive
* Male sex (subjects providing and/or testing human semen specimens)
* For males providing human semen specimens, either healthy subjects or men receiving health care for any one or more of the following reasons:

  * Partner in a couple having difficulty conceiving
  * Diagnosed with male factor infertility
  * Post-vasectomy patients
  * Post-vasectomy reversal patients

Testers Only

* Be able to provide signed Informed Consent
* 20 - 50 years of age inclusive

Exclusion Criteria:

* Any medical or personal issue that would impair the ability of the subject to adhere to the protocol (e.g. substance abuse, neurological disorders)
* Patients currently taking investigational drugs or who are active participants in a treatment trial for any condition
* Unable to speak, understand, or write English
* Mental illness that would interfere with understanding during the discussion of Informed Consent or that would compromise ability to follow the study protocol including, but not limited to, review of the TRAK™ Instructional Booklet, semen specimen collection, and semen specimen testing.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 272 (Actual)
Dates: Start 2015-09-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Dula, MD, Principal Investigator — San Fernando Valley Urological Associates Medical Group; Robert Boostanfar, MD, Principal Investigator — California Reproductive Services: Huntington Reproductive Center
Locations (3):
- United States (3):
  - California Reproductive Services: Huntington Reproductive Center, Encino, California
  - San Fernando Valley Urological Associates Medical Group, Tarzana, California
  - Men's Fertility Laboratory, Great Neck, New York

REFERENCES:
- [Derived] Schaff UY, Fredriksen LL, Epperson JG, Quebral TR, Naab S, Sarno MJ, Eisenberg ML, Sommer GJ. Novel centrifugal technology for measuring sperm concentration in the home. Fertil Steril. 2017 Feb;107(2):358-364.e4. doi: 10.1016/j.fertnstert.2016.10.025. Epub 2016 Nov 22. PMID 27887718

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men were recruited at three medical clinic sites from 2 September 2015 to 4 December 2015.
Groups:
- Donor/Tester Subjects: Male subjects use the TRAK device to attain a measurement of sperm concentration from a semen specimen
  TRAK device: Use of TRAK to attain sperm concentration measurement
- Tester Only Subjects: Male or female subjects use the TRAK device to attain a measurement of sperm concentration from a semen specimen
  TRAK device: Use of TRAK to attain sperm concentration measurement
Period: Overall Study
Arm/Group | Donor/Tester Subjects | Tester Only Subjects
Started | 258 | 14
Completed | 228 | 11
Not Completed | 30 | 3
Not completed — Protocol Violation | 30 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donor/Tester Subjects | Tester Only Subjects | Total
Number analyzed (Participants) | 258 | 14 | 272
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 258 | 14 | 272
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [27 to 40] | 33 [27.5 to 35.5] | 34 [27 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 14 | 14
  Male | 258 | 0 | 258
Region of Enrollment [Number; unit: participants]
  United States | 258 | 14 | 272

OUTCOME MEASURES:

1. Primary Outcome: Number of Untrained Lay Users That Obtained Accurate and Inaccurate Subfertility Results From the TRAK Device When Compared to Results Obtained From the Gold Standard
Description: Lay users obtained categorical sperm concentration result. Positive (for subfertility) results are less than or equal to 15 M/mL threshold. Gold standard reference (analysis by Computer-aided Semen Analysis [CASA]) result was measured and compared to Trak. True positive and true negative matched Reference category result and false negative, false positive did not match gold standard reference category result.
Time Frame: Participants will be followed for one visit for up to 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Donor/Tester Subjects | Tester Only Subjects
Number analyzed (Participants) | 228 | 11
Participants
  True Positive Trak Results | 52 | 2
  True Negative Trak Results | 160 | 7
  False Positive Trak Results | 10 | 2
  False Negative Trak Results | 6 | 0
Statistical Analysis 1: Comparison: Donor/Tester Subjects vs Tester Only Subjects; Test type: Other; Sensitivity = 90.0, 95% CI 2-sided [79.9 to 95.3] — Sensitivity estimates the percent true positive results obtained by Trak. Positive results are less than 15 M/mL sperm concentration and are part of a sub fertile diagnostic assessment
Statistical Analysis 2: Comparison: Donor/Tester Subjects vs Tester Only Subjects; Test type: Other; Specificity = 93.3, 95% CI 2-sided [88.7 to 96.1] — Specificity is calculated by the percentage of true negative results obtained using Trak compared to reference method. Negative (for subfertility) results are greater than 15 M/mL

2. Secondary Outcome: Number of Accurate and Inaccurate Subfertility Results as Obtained by Healthcare Professionals Observing Assays Result Performed by Untrained Lay Users.
Description: Healthcare professions obtained a categorical sperm concentration result by observing completed assay outputs as performed by Lay Users. Positive (for subfertility) results are less than or equal to 15 M/mL threshold. Reference result using gold standard (CASA) was measured and compared to Trak. True positive and true negative matched Reference category result and false negative, false positive did not match reference category result.
Time Frame: Participants will be followed for one visit for up to 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Donor/Tester Subjects | Tester Only Subjects
Number analyzed (Participants) | 228 | 11
Participants
  True Positive Trak Results | 56 | 1
  True Negative Trak Results | 161 | 7
  False Positive Trak Results | 9 | 2
  False Negative Trak Results | 2 | 1
Statistical Analysis 1: Comparison: Donor/Tester Subjects vs Tester Only Subjects; Test type: Other; Sensitivity = 95.0, 95% CI 2-sided [86.3 to 98.3]
Statistical Analysis 2: Comparison: Donor/Tester Subjects vs Tester Only Subjects; Test type: Other; Specificity = 94.9, 95% CI 2-sided [90.6 to 97.3]

3. Secondary Outcome: Number of Accurate and Inaccurate Results Obtained by Healthcare Professionals Performing Trak Assays on Subjects' Samples.
Description: Healthcare professions obtained a categorical sperm concentration result by performing assay on aliquot obtained from Lay User's sample. Positive (for subfertility) results are less than or equal to 15 M/mL threshold. Reference result using gold standard (CASA) was measured and compared to Trak. True positive and true negative matched Reference category result and false negative, false positive did not match reference category result.
Time Frame: Participants will be followed for one visit for up to 2 hours
Population: One fewer was analyzed in this population because a sample did not have enough sample to allow the HCP to run the test.
Measure: Count of Participants; unit: Participants
Arm/Group | Donor/Tester Subjects | Tester Only Subjects
Number analyzed (Participants) | 227 | 11
Participants
  True Positive Trak Results | 57 | 1
  True Negative Trak Results | 160 | 7
  False Positive Trak Results | 9 | 2
  False Negative Trak Results | 1 | 1
Statistical Analysis 1: Comparison: Donor/Tester Subjects vs Tester Only Subjects; Test type: Other; Sensitivity = 96.7, 95% CI 2-sided [88.7 to 99.1]
Statistical Analysis 2: Comparison: Donor/Tester Subjects vs Tester Only Subjects; Test type: Other; Specificity = 93.8, 95% CI 2-sided [89.2 to 96.5]

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | Donor/Tester Subjects | Tester Only Subjects
Serious Adverse Events (participants affected / at risk) | 0/258 | 0/14
Other Adverse Events (participants affected / at risk) | 0/258 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No